CLINICAL TRIAL: NCT06247735
Title: A Phase 2, Randomized, Placebo-controlled, Parallel Group, Multicenter 12-week Study With a 52-week Extension to Evaluate the Efficacy and Safety of Two Doses of K-808 (Pemafibrate) in Subjects With Primary Biliary Cholangitis With Inadequate Response to Ursodeoxycholic Acid and/or Obeticholic Acid Treatment
Brief Title: Study to Evaluate the Efficacy and Safety of K-808 (Pemafibrate) in Participants With Primary Biliary Cholangitis (PBC) With Inadequate Response to Ursodeoxycholic Acid (UDCA) and/or Obeticholic Acid (OCA) Treatment.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-808-2.01
Record Dates: First submitted 2024-01-22; First posted 2024-02-08 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — (R)-2-(3-((benzoxazol-2-yl-d4 (3-(4-methoxyphenoxy-d7)propyl)amino)methyl)phenoxy) butanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo + K-877 (Group A) (Placebo Comparator): Placebo for 12 Weeks followed by K-808 (Dose A) for 52 Weeks
  Interventions: Drug: K-808 (Dose A); Drug: Placebo
- Placebo + K-877 (Group B) (Placebo Comparator): Placebo for 12 Weeks followed by K-808 (Dose B) for 52 Weeks
  Interventions: Drug: K-808 (Dose B); Drug: Placebo
- K-808 Group A (Experimental): K-808 (Dose A) for 64 Weeks
  Interventions: Drug: K-808 (Dose A)
- K-808 Group B (Experimental): K-808 (Dose B) for 64 Weeks
  Interventions: Drug: K-808 (Dose B)

INTERVENTIONS:
Drug: K-808 (Dose A) — Administered orally once daily
  Other Names: Pemafibrate
  Arms: K-808 Group A; Placebo + K-877 (Group A)
Drug: K-808 (Dose B) — Administered orally once daily
  Other Names: Pemafibrate
  Arms: K-808 Group B; Placebo + K-877 (Group B)
Drug: Placebo — Administered orally once daily
  Arms: Placebo + K-877 (Group A); Placebo + K-877 (Group B)

SUMMARY:
Study to investigate the efficacy and safety of two doses of K-808 (pemafribate) in subjects with PBC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant who has a PBC diagnosis as demonstrated by the presence of ≥2 of the following three diagnostic criteria:

  * History of ALP above ULN for at least 6 months
  * History of positive antimitochondrial antibody (AMA) titer or positive PBC-specific antinuclear antibody (ANA) titer
  * Historical liver biopsy consistent with PBC
* Participant has the following qualifying biochemistry value at Screening:

  * ALP ≥1.5 × ULN
* Participant is ≥18 years of age at consent.
* Participant meets all other eligibility criteria outlined in the Clinical Study Protocol.

Exclusion Criteria:

* Participant meets any one of the following criteria at Screening:

  * ALP>10 × ULN
  * ALT or AST >5 × ULN
  * Hepatitis C treatment within 5 years of Screening, or active hepatitis C as defined by positive hepatitis C antibody with the presence of hepatitis C virus ribonucleic acid; subjects with active hepatitis B (HBV) infection (hepatitis B surface antigen [HbsAg] positive) will be excluded. A subject with resolved hepatitis A at least 3 months prior to the Screening Visit can be screened.
  * Primary sclerosing cholangitis and secondary sclerosing cholangitis (eg, due to cholangiolithiasis, ischemia, telangiectasia, vasculitis, infectious diseases)
  * Alcoholic liver disease
  * History of definite autoimmune hepatitis or PBC/autoimmune hepatitis overlap, defined as both of the following: 1) IgG >2 × ULN and/or positive anti-smooth muscle antibodies, 2) liver histology revealing moderate or severe periportal or periseptal inflammation
  * Nonalcoholic steatohepatitis (NASH)
  * Gilbert's Syndrome
  * Alpha-1-antitrypsin deficiency, cystic fibrosis, Wilson's disease, hemochromatosis based on historically established diagnosis
  * Drug-induced liver injury (DILI) as defined by typical exposure and history
  * Known condition that involves bile duct obstruction or cholestasis other than PBC, eg, vascular diseases (eg, Budd-Chiari syndrome, sinusoidal obstruction syndrome, congestive hepatopathy), congenital conditions (ductal plate malformations, Caroli syndrome, congenital liver fibrosis), idiopathic ductopenia
  * Hepatocellular carcinoma
* Participant meets any other exclusion criteria outlined in the Clinical Study Protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in serum alkaline phosphatase (ALP) | Baseline to Week 12
  Two doses of K-808 compared to placebo after 12 weeks of treatment

SECONDARY OUTCOMES:
Achievement of normalization of ALP level | Baseline to Week 12
  ALP ≤1 × upper limit of normal (ULN)
Achievement of target levels of ALP and total bilirubin (TB) | Baseline to Weeks 12 and 64
  After two doses of K-808
Change from baseline in liver function parameters | Baseline to Weeks 12 and 64
  liver function test results including ALP, total and conjugated bilirubin, albumin, international normalized ratio [INR], γ-GT, ALT, AST, albumin, platelets count
Change from baseline in GLOBE risk score | Baseline to Weeks 12 and 64
  calculated by GLOBE scoring system which is calculated based on serum values of bilirubin, ALP, albumin and platelet count.
Change from baseline in UK-PBC score | Baseline to Weeks 12 and 64
  PBC risk score developed by United Kingdom (UK)-PBC Consortium is a scoring system and the calculation is based on laboratory test measurements and upper limits of normal (ULN) for the total bilirubin (BIL12); alanine transaminase or aspartate transaminase (TA12), and alkaline phosphatase (ALP12) after at least 12 months of UDCA, and the laboratory test measurements and lower limits of normal (LLN) for the serum albumin and platelet count in the same timeframe. A high number is indicative of a worse score.
Incidence of Treatment Emergent Adverse Events (TEAEs) | Baseline to Week 68
  Coded using the most recent version of Medical Dictionary of Regulatory Activities (MedDRA).

CONTACTS AND LOCATIONS:
Overall Officials: Andre Belous, MD, PhD, Study Director — Kowa Pharma Development Co.
Locations (38):
- United States (21):
  - UA Thomas D. Boyer Liver Institute, Tucson, Arizona
  - Southern California Research Center - Coronado, Coronado, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Velocity Clinical Research, Santa Ana, California
  - Peak Gastroenterology Associates Colorado Springs, Colorado Springs, Colorado
  - University of Florida Hepatology Research at CTRB, Gainesville, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - University of Miami Leonard M. Miller School of Medicine, Miami, Florida
  - Springfield Clinic, Springfield, Illinois
  - Mercy Medical Center - Mcauley Plaza, Baltimore, Maryland
  - CommonSpirit Health Research Institute, Omaha, Nebraska
  - New York University Hepatology Associates, New York, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Rapid City Medical Center, Rapid City, South Dakota
  - Vanderbilt Digestive Disease Center, Nashville, Tennessee
  - Pioneer Research Solutions, Houston, Texas
  - UVA Health - University of Virginia Health System, Charlottesville, Virginia
  - Gastrointestinal and Liver Specialists of Tidewater - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Liver Institute Northwest, Seattle, Washington
- Canada (4):
  - (G.I,R,I) GI Research Institute, Vancouver, British Columbia
  - Office of Dr. Gauthier, North Bay, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Centre de Recherche du Centre Hospitalier de l'Université de Montréal (CRCHUM), Montreal, Quebec
- Japan (13):
  - 306, Fukui
  - 313, Fukuoka
  - 305, Hamamatsu
  - 308, Hirakata
  - 309, Hiroshima
  - 304, Isehara
  - 303, Itabashi-ku
  - 312, Kanazawa
  - 307, Matsumoto
  - 311, Ōmura
  - 302, Sapporo
  - Teine Keijinkai Hospital, Sapporo
  - 314, Yokohama

IPD SHARING:
Plan to Share IPD: Yes